CLINICAL TRIAL: NCT05795907
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Ascending Single and 14-day Repeated Oral Doses of SAR443820 in Healthy Adult Participants.
Brief Title: Single & Multiple Ascending Dose Study of SAR443820 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TDU16519-TDR16520; U1111-1254-0034 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis (Healthy Volunteers)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Part 1b with open label study design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAR443820 (Experimental): Single dose oral ascending dose (parts 1a and 1b) and multiple ascending oral dose (part 2) of SAR443820
  Interventions: Drug: SAR443820
- Placebo (Placebo Comparator): Single dose oral ascending dose (part 1a) and multiple ascending oral dose (part 2) of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR443820 — Capsule / Oral
  Arms: SAR443820
Drug: Placebo — Matching Capsule / Oral
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-center study conducted in 2 parts:

Part 1a, single ascending dose (SAD-TDU16519): Double-blind, randomized, placebo-controlled sequential ascending single oral doses including up to 6 cohorts. Each cohort will include 8 participants (6 receiving SAR443820 and 2 placebo).

Part 1b (TDU16519): - Open label, single SAR443820 dose in one or two separated cohort(s) for SAR443820 measurements in CSF and in plasma.

Part 2, multiple ascending dose (MAD -TDR16520): Double-blind, randomized, placebo-controlled, sequential ascending repeated oral doses for 14 days, including up to 4 cohorts. Each cohort will include 10 participants (8 receiving SAR443820 and 2 placebo).

DETAILED DESCRIPTION:
The duration of the study for a participant will include:

Screening Period: up to 28 days

Part 1a:

Treatment in fasted condition: 1 day (Day 1). Study observation Period from Day -2/Day -1 to Day 3. Follow-up with the end of study: from Day 5 to Day 7. Total duration from screening per participant: up to 5 weeks.

Part 1b:

Treatment in fed condition: 1 day (Day 1). Study observation Period from Day -1/Day1 to Day 2. Follow-up with the end of study: from Day 5 to Day 7. Total duration from screening per participant: up to 5 weeks.

Part 2:

Treatment: 14 days (Day 1 to Day 14). Study observation Period from Day -2/Day -1 to Day 17. Follow-up with the end of study: from Day 19 to Day 21. Total duration from screening per participant: up to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

Male and/or female participant, between 18 and 55 years of age, inclusive. Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m2, inclusive.

Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).

Having given written informed consent prior to undertaking any study-related procedure.

Not under any administrative or legal supervision or under institutionalization due to regulatory or juridical order.

Exclusion Criteria:

Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteo-muscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness.

Personal medical history of seizure.

Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).

Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.

Positive result for hepatitis B, C or HIV

Positive result on urine drug screen

Positive alcohol test.

Any consumption of citrus fruits or their juices within 5 days before inclusion.

Current psychiatric disorder, suicidal ideation in the previous 6 months (as assessed by the C-SSRS), or a lifetime suicide attempt.

Additional exclusion criteria applied, and specially for Part 1b, criteria related to the study procedure of lumbar puncture.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Parts 1a and 1b: Number of participants with adverse events | Day1 up to Day 7 (end of study visit)
Part 2: Number of participants with adverse events | Day1 up to Day 21 (end of study visit)

SECONDARY OUTCOMES:
Parts 1a and 1b: Assessment of pharmacokinetic parameter of SAR443820: Cmax in plasma | Day1
  Parts 1a and 1b: Maximum plasma concentration
Parts 1a and 1b: Assessment of pharmacokinetic parameter of SAR443820: tmax in plasma | Day 1
  Parts 1a and 1b: time to reach Cmax
Parts 1a and 1b : Assessment of pharmacokinetic parameter of SAR443820: AUC in plasma | Day1
  Parts 1a and 1b: Area under the plasma concentration versus time
Parts 1a and 1b : Assessment of pharmacokinetic parameter of SAR443820: t1/2z in plasma | Day1
  Terminal half-life in plasma
Part1b: SAR443820 concentrations in cerebrospinal fluid (CSF) samples | Day1
  Part 1b: CSF to plasma concentration ratio
Part 2: Assessment of pharmacokinetic parameter of SAR443820: Cmax in plasma | Day1 and Day14
  Part 2: Maximum plasma concentration
Part 2: Assessment of pharmacokinetic parameter of SAR443820: tmax in plasma | Day1 and Day14
  Part 2: Time to reach Cmax
Part 2: Assessment of pharmacokinetic parameter of SAR443820: AUC tau in plasma | Day1 and Day14
  Part 2: Area under the plasma concentration versus time during a dosing interval
Part 2 Assessment of pharmacokinetic parameter of SAR443820: t1/2z in plasma | Day14
  Terminal half-life in plasma
Part 2: Day14/Day1 of 4β-hydroxycholesterol ratio in plasma | Day1 and Day14
  D14/D1 of 4β-hydroxycholesterol ratio

CONTACTS AND LOCATIONS:
Overall Officials: Trial Transparency email recommended (Toll free for US & Canada), Study Director — Sanofi; Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Prism Research-Site Number:8400001, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Hincelin-Mery A, Nicolas X, Cantalloube C, Pomponio R, Lewanczyk P, Benamor M, Ofengeim D, Krupka E, Hsiao-Nakamoto J, Eastenson A, Atassi N. Safety, pharmacokinetics, and target engagement of a brain penetrant RIPK1 inhibitor, SAR443820 (DNL788), in healthy adult participants. Clin Transl Sci. 2024 Jan;17(1):e13690. doi: 10.1111/cts.13690. Epub 2023 Dec 11. PMID 38010108